CLINICAL TRIAL: NCT02072499
Title: The Effect of KTP (Potassium-titanyl-phosphate) Green Light Prostatectomy (180W) Compared With Open Prostatectomy When Treating Benign Prostatic Hyperplasia, a Prospective Randomized Study
Brief Title: KTP Green Light Prostatectomy Compared With Open Prostatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Hannu Koistinen, MD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 164/13/03/02/08
Record Dates: First submitted 2013-12-17; First posted 2014-02-26 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- KTP Green Light Prostatectomy (Experimental): Device
  Interventions: Procedure: KTP Green Light Prostatectomy; Device: Green Light
- Open prostatectomy (Active Comparator): Surgical procedure
  Interventions: Procedure: Open prostatectomy

INTERVENTIONS:
Procedure: KTP Green Light Prostatectomy
  Arms: KTP Green Light Prostatectomy
Device: Green Light
  Arms: KTP Green Light Prostatectomy
Procedure: Open prostatectomy
  Arms: Open prostatectomy

SUMMARY:
The purpose of this study is to compare safety and efficacy of Green Light PVP (Photoselective Vaporisation of the Prostate) compared to open prostatectomy when treating benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing surgery for BPH with prostate size more than 100cc

Exclusion Criteria:

* Previous prostate surgery
* Carcinoma of the prostate
* Neurogenic bladder
* Bladder carcinoma

Ages: 40 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2017-06 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
IPSS (International Prostate Symptom Score) | 12 months
  symptom score

SECONDARY OUTCOMES:
DAN-PSS (Danish Prostate Symptom Score) | 0, 3, 6 and 12 months
  symptom score
Maximum flow rate (Qmax) | 0, 3, 6 and 12 months
Residual urine | 0, 3, 6 and 12 months
Length of catheterization | Participants will be followed for the duration of hospital stay, an expected maximum of two weeks
Length of hospital stay | Participants will be followed for the duration of hospital stay, an expected maximum of two weeks
Perioperative bleeding | Time of operation
IIEF (International Index of Erectile Function questionnaire) | 0,12 months
Prostate volume measured with TRUS (transrectal ultrasound) | 0, 12 moths
Rate of unscheduled hospital contacts | 12 months
IPSS (International Prostate Symptom Score) | 0, 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland